CLINICAL TRIAL: NCT07135453
Title: Novel Serotype Alert: Investigate New Pneumococcal Conjugate Vaccines for Inducing Cross-protection Against Newly Discovered Serotype 33E and Putative Novel Serogroup 33 Serotypes
Brief Title: Induction of Cross-protective Antibodies for Serogroup 33 by Pneumococcal Conjugate Vaccines
Acronym: Group 33/PCVs
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, David Lafon, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300008528(000544386); MISP102547 (Other Grant/Funding Number: Merck Corporation)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-08

CONDITIONS: Vaccine; Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PCV20 (Experimental): Will receive PCV20
  Interventions: Biological: Pneumococcal Vaccine
- PCV21 (Experimental): Will receive PCV21
  Interventions: Biological: Pneumococcal Vaccine

INTERVENTIONS:
Biological: Pneumococcal Vaccine — PCV

SUMMARY:
The goal of this study is to learn whether different types of vaccines to prevent bacterial infections are able to effectively create antibodies that defend against certain types of bacteria.

We will give two different types of vaccine and evaluate the effectiveness of antibodies produced by each vaccine in killing bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult

Exclusion Criteria:

* No prior history of pneumococcal vaccination
* No immunosuppressing medications or chronic diseases that affect immune function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Serogroup 33 antibodies | 4 weeks post-vaccination
  Serum antipneumococcal antibody concentrations (micrograms/mL) against members of serogroup 33, measured using WHO-ELISA
Antibody-mediated killing | 4 weeks post-vaccination
  Opsonic activity of vaccine-induced antibodies (reported as opsonic index, or OI); measured using an opsonophagocytic killing (OPK) assay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided